CLINICAL TRIAL: NCT02027857
Title: Comparison of the Application in Traumatic Brain Edema Between Electrical Impedance Tomography and Non-invasive Intracranial Pressure Monitoring
Brief Title: Comparison of the Application in Traumatic Brain Edema Between EIT and Non-invasive ICP Monitoring
Acronym: EIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 20131211-8
Record Dates: First submitted 2013-12-23; First posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Brain Electrical Impedance;; Non-invasive Intracranial Pressure
Keywords: brain electrical impedance;; traumatic brain injury;; brain edema;; intracranial pressure
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- mannitol empirical therapy (No Intervention): There would be 20 patients in this group, who would be given mannitol to relieve the brain edema depending on the empirical therapy by doctors.
- EIT monitoring (Experimental): There would be 20 patients in this group, who would be given mannitol to relieve the brain edema depending on the results of Electrical impedance tomography monitoring.
  Interventions: Device: EIT monitoring
- non-invasive ICP monitoring (Other): There would be 20 patients in this group, who would be given mannitol to relieve the brain edema depending on the results of non-invasive intracranial pressure monitoring.
  Interventions: Device: non-invasive ICP monitoring

INTERVENTIONS:
Device: EIT monitoring
  Arms: EIT monitoring
Device: non-invasive ICP monitoring
  Arms: non-invasive ICP monitoring

SUMMARY:
Brain edema is the main reason for the disability and lethality in traumatic brain injury, which is the most difficult part of emergency rescue. Recently, there is no medical equipment to monitor the early brain edema in clinic. We have found that Electrical impedance tomography (EIT) can perform the real-time and bedside monitoring of brain electrical impedance after single-dose mannitol treatment, which may be a new strategy for the surveillance of brain edema. In this study, we would like to compare the application in traumatic brain edema between EIT and Noninvasive intracranial pressure (ICP) monitoring, including the progress of brain edema, the relationship between impedance and ICP, and the improvement for the patients' prognosis. EIT would probably be a new image strategy for the treatment of traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients were 16 to 65 years of age with all genders.
2. The patients had been diagnosed as traumatic brain injury during 24 hours before enrollment, with the confirmation of CT or MRI.
3. All the patients had provided written informed consent.

6. The patients were receiving usual inpatient rehabilitation and conservative treatment .

Exclusion Criteria:

1. The patients with indication of operation during the research should be excluded.
2. The patients were assessed as unqualified for the study according to the comprehensive evaluation opinion brought forward by the research team.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
brain electrical impedance | From the 1st day (enrollment) to the 7th day
  After the patients' enrollment, the electrodes would be placed properly and the continuous monitoring of brain impedance just be started.

SECONDARY OUTCOMES:
Glasgow coma scale(GCS) | on the 0 day of the study
  The scale is composed of three tests: eye, verbal and motor responses. The three values separately as well as their sum are considered. The lowest possible GCS (the sum) is 3 (deep coma or death), while the highest is 15 (fully awake person).
demographic characteristics at baseline | on the 0 day of the study
  The demographic data include age, gender, injuries reason, time from injuries, and so on.
kidney function examination | On the 1st day, 3rd day, 5th and 7th day
  There are three main indicators: blood creatinine, urea nitrogen, and uric acid. These indicator are used as a monitor of the kidney safety.
Physiological and pathological reflex check | on the 1st and 7th day
muscular strength and tension test | on the 1st and 7th day
  There are 6 grades in muscular strength test. And muscular tension test was referred to Modified Ashworth scale.
non-invasive intracranial pressure | From the 1st day (enrollment) to the 7th day
  This equipment can continuously monitor the change of intracranial pressure since the patients' enrollment.
brain CT scan | On the 1st day (enrollment), and 7th day
  Brain CT scan is applied to monitor the degree and progress of the brain change after the medication of mannitol.
Disability Rating Scale (DRS) | on the 1st day (enrollment), seventh day after hospitalization
  The DRS includes measures of eye opening, verbalization, and motor response (derived from the Glasgow Coma Scale); cognitive understanding of feeding, dressing, and grooming; degree of assistance and supervision required; and employability. Scores range from 0 to 29, with higher values indicating greater disability.
glasgow outcome scale(GOS) | the patients were discharged or the 7th day after hospitalization
  GOS includes 5 grades: Dead, Vegetative state, Severe disability, Moderate disability, Good recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Zhou, M.D.; Ph.D., Study Director — Department of Neurosurgery, Xijing Hospital, Fourth Military Medical University
Locations (1):
- Department of Neurosurgery, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China